CLINICAL TRIAL: NCT04716569
Title: Faculty of Medicine ,South Valley University
Brief Title: Evaluation of Ivermectin Mucoadhesive Nanosuspension as Nasal Spray in Management of Early Covid-19
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: South Valley University (Other)
Responsible Party: Principal Investigator, Zaky Aref, ass.professor, South Valley University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SVU MED CIT0 23 4 21 1 120
Record Dates: First submitted 2021-01-19; First posted 2021-01-20 (Actual); Last update posted 2021-03-17 (Actual); Status verified 2021-03

CONDITIONS: Covid19
Keywords: Ivermectin intranasal spray in covid19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- intranasal Ivermectin group (Experimental): Ivermectin group Patients who will receive intranasal ivermectin
  Interventions: Drug: intranasal ivermectin spray
- Control group (Other): patients who will receive regular protocol drugs
  Interventions: Drug: intranasal ivermectin spray

INTERVENTIONS:
Drug: intranasal ivermectin spray — usage of ivermectin as intranasal spray for treating early covid patiens

SUMMARY:
Ivermectin showed a strong viricidal effect upon covid19 virus in vitro as proved by many authors according to many studies , covid virus stay in postnasal space for 4 days before starting general manifestation, so ivermectin mucoadhesive nanosuspension sprayed inside the nose and post nasal space may help in early management of covid19 and may play a great rule in prophylaxis as well

DETAILED DESCRIPTION:
150 patient with early covid is devided into two groups first group will receive regular protocol of drugs second group will receive ivermectin nasal spray in addition to regular protocl of drugs

ELIGIBILITY:
Inclusion Criteria:

* early covid19 pateints

Exclusion Criteria:

* children and pregnant women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2021-01-20 (Actual); Primary Completion 2021-02-20 (Actual); Study Completion 2021-03-20 (Estimated)

PRIMARY OUTCOMES:
progression of covid 19 clinical picture | [ Time Frame: within 14 days after enrollement ]
  progress of Symptoms ( Fever ,Cough, Sore Throat, Myalgia,Diarrhea, Shortness of Breath)with radiological assesment and blood tests

CONTACTS AND LOCATIONS:
Locations (1):
- Zaky Aref, Qina, Qena Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Aref ZF, Bazeed SEES, Hassan MH, Hassan AS, Rashad A, Hassan RG, Abdelmaksoud AA. Clinical, Biochemical and Molecular Evaluations of Ivermectin Mucoadhesive Nanosuspension Nasal Spray in Reducing Upper Respiratory Symptoms of Mild COVID-19. Int J Nanomedicine. 2021 Jun 15;16:4063-4072. doi: 10.2147/IJN.S313093. eCollection 2021. PMID 34163159